CLINICAL TRIAL: NCT00621478
Title: Use Of Lorazepam For The Treatment Of Pediatric Status Epilepticus: A Randomized, Double-Blinded Trial Of Lorazepam And Diazepam
Brief Title: Efficacy and Safety Study Comparing Lorazepam and Diazepam for Children in the Emergency Department With Seizures (Status 2)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01HD043393; 275200403393C
Record Dates: First submitted 2008-02-20; First posted 2008-02-22 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-07

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Lorazepam; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Active Comparator): Cohort 1 (preconsented) patients will involve obtaining informed consent from the legally authorized representative of a potential study subject before they present to the ED in SE. Patient assent will be obtained for patients as per local IRB rules. The consent document (enclosed in this application) will inform parents that if their child comes to the ED and qualifies for the study based on study inclusion/exclusion criteria, they will be enrolled.
  Patients who cannot be contacted to confirm consent will be enrolled in Cohort 2 (EFIC) as detailed below.
  Patients in Cohort 1 will be randomized in a blinded fashion to either lorazepam 0.1 mg/kg or diazepam 0.2 mg/kg
  Interventions: Drug: lorazepam or diazepam
- Cohort 2 (Active Comparator): Cohort 2 (EFIC) will include patients who appear in the ED with SE and qualify for the study but have not given prior consent. These patients will be enrolled under the EFIC regulations. The parent/guardian will be given the opportunity to object to participation or ask additional questions.
  The child will be enrolled (dosed) with study medication under an EFIC. Once the child is stabilized, a research staff member will approach the parent or LAR to obtain informed consent to continue the child's participation in the study. If a parent or LAR refuses continued participation, then no further study procedures will be performed. Safety and data will be collected in accordance with federal regulations.
  Cohort 2 will be randomized, like Cohort 1, to either lorazepam 0.1 mg/kg or diazepam 0.2 mg/kg
  Interventions: Drug: lorazepam or diazepam

INTERVENTIONS:
Drug: lorazepam or diazepam — Administration instructions will ask to deliver 0.04 ml per kilogram of child's weight of the study medication up to a maximum of 1.6 ml. 0.04 ml/kg (maximum dose 1.6 ml) will deliver 0.1 mg/kg of lorazepam (maximum dose 4 mg) and 0.2 mg/kg of diazepam (maximum dose 8 mg). Half of this dose can be repeated in 5 minutes if the patient is still convulsing.
  The medication will be administered as a slow IV push.
  Other Names: Ativan; Valium

SUMMARY:
Children with seizures are frequently seen in the emergency department. The drug lorazepam, which is commonly used, is not labeled by the US Food and Drug Administration for children for this use. The FDA, under the Best Pharmaceuticals for Children Act, has requested that a study comparing diazepam, a drug that is labeled by the FDA for this indication, with lorazepam be performed. The study will show whether one drug is more effective and safe than the other.

DETAILED DESCRIPTION:
Textbooks and expert opinion recommend both diazepam and lorazepam as initial therapy for children in status epilepticus (SE) and provide recommended doses that are commonly used. However, unlike diazepam, lorazepam is only FDA-approved for treatment for SE in patients over 18 years of age. Despite this fact, many experts support the use of lorazepam over diazepam in pediatric SE. Increased duration of action, increased effectiveness in terminating SE, and a lower incidence of respiratory depression have been cited as potential advantages of lorazepam over diazepam. However, data to support firm recommendations for one medication over another are lacking. Thus, either diazepam (FDA-approved) or lorazepam can be considered first-line agents for pediatric SE, and the physician's choice of agent depends on local practice patterns and individual treatment styles. In the prehospital (Emergency Medical Services) setting, diazepam is commonly chosen because of a longer shelf life without refrigeration.

The purpose of this study is to determine the differences in efficacy and safety between these two commonly used benzodiazepines, as requested by the FDA under the Best Pharmaceuticals for Children Act, using the Exception from Informed Consent provided by the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 months to less than 18 years;
2. Generalized tonic clonic status epilepticus, defined as:

   1. Three or more generalized tonic clonic seizures within the last hour and currently experiencing a convulsion (i.e. the current convulsion may be the third convulsion within one hour); or
   2. Two or more generalized tonic clonic seizures in succession with no recovery of consciousness between seizures and currently experiencing a convulsion (i.e. the current convulsion may be the second convulsion without recovery of consciousness after the first convulsion); or
   3. A seizure that lasts at least 5 minutes that is either generalized tonic clonic in its entirety or starts focal and then generalizes. The seizure must be associated with loss of consciousness

Exclusion Criteria:

1. Pregnancy;
2. Shock prior to study drug (sustained hypotension requiring inotropic therapy);
3. Significant dysrhythmia prior to study drug (other than sinus tachycardia);
4. Need for emergent surgical intervention and general anesthesia for a condition present prior to study drug;
5. Known sensitivity to benzodiazepines or known contraindication to benzodiazepine use; or
6. Use of a benzodiazepine within 1 week of presentation.

Certain exclusion criteria may not be known at the time of drug administration due to the need for emergent treatment. Thus patients will be terminated from the study (early terminators) if the investigators discover any of the following conditions after administration of study drug:

1. Pregnancy;
2. Use of a benzodiazepine within 1 week of presentation.
3. Parent/guardian refusal to give informed consent by the methods described;
4. Patient's refusal to assent (for patients ≥ 7 yrs old and mentally competent to understand study procedures) by the methods described, or as required by the local IRB;

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 259 (Actual)
Dates: Start 2008-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
cessation of convulsions within 10 minutes of the initial administration of the study drug and a sustained absence of convulsions for 30 minutes from the initial administration of the study drug. | 30 minutes

SECONDARY OUTCOMES:
To determine population pharmacokinetics (PK) of lorazepam using sparse sampling. | 24 hr
feasibility of identifying patients for informed consent prior to arrival in status epilepticus for a randomized controlled trial | 2 years
the experience of community consultation and public disclosure | 2 years
feasibility of enrolling pediatric patients under an exception from informed consent | 2 years
determine patients' and parents' attitudes and reactions to an exception from informed consent approach | 2 years
severe or life-threatening respiratory depression | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: James Chamberlain, MD, Principal Investigator — Children's National Research Institute
Locations (14):
- United States (12):
  - University of California- Davis Medical Center, Davis, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Maryland Hospital for Children, Baltimore, Maryland
  - University of Michigan Emergency Medicine Research, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital of Buffalo, Buffalo, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah Pediatric Emergency Medicine, Salt Lake City, Utah
  - Medical College of Wisconsin Children's Corporate Center, Milwaukee, Wisconsin
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

REFERENCES:
- [Derived] Chamberlain DB, Chamberlain JM. Making Sense of a Negative Clinical Trial Result: A Bayesian Analysis of a Clinical Trial of Lorazepam and Diazepam for Pediatric Status Epilepticus. Ann Emerg Med. 2017 Jan;69(1):117-124. doi: 10.1016/j.annemergmed.2016.08.449. PMID 27993298
- [Derived] Chamberlain JM, Okada P, Holsti M, Mahajan P, Brown KM, Vance C, Gonzalez V, Lichenstein R, Stanley R, Brousseau DC, Grubenhoff J, Zemek R, Johnson DW, Clemons TE, Baren J; Pediatric Emergency Care Applied Research Network (PECARN). Lorazepam vs diazepam for pediatric status epilepticus: a randomized clinical trial. JAMA. 2014 Apr 23-30;311(16):1652-60. doi: 10.1001/jama.2014.2625. PMID 24756515